CLINICAL TRIAL: NCT03554343
Title: Sun May Arise on SMA : Newborn Screening of SMA in Belgium
Brief Title: Sun May Arise on SMA : Newborn Screening of Spinal Muscular Atrophy in Belgium
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional de la Citadelle (Other)
Collaborators: AveXis, Inc. (Industry); Biogen (Industry); Roche Pharma AG (Industry); Association Belge contre les Maladies neuro Musculaires (Unknown)
Responsible Party: Principal Investigator, Laurent Servais, Professor, Centre Hospitalier Régional de la Citadelle
Other Study IDs: B412201734396
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: newborn screening
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA is exctracted from the Guthrie Dried Blood Test Analysis is performed by the genetic department of Liege University Hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All newborn from Southern Belgium: All newborns except newborns for which parents refuse newborn screening will be tested for exon 7 deletion in survival motor neuron 1 (SMN1)
  Interventions: Diagnostic Test: test for SMN1 exon 7 deletion

INTERVENTIONS:
Diagnostic Test: test for SMN1 exon 7 deletion — Newborns are screened for SMN1 exon 7 deletion through standard NBS practice Positive case are promptly referred to reference centers

SUMMARY:
Medico-economic study of Newborn screening of Spinal Muscular Atrophy

DETAILED DESCRIPTION:
The aim of this project is to demonstrate the feasibility and the medico-economic impact of a spinal muscular atrophy neonatal screening in a European country. We propose a 3-year-neonatal screening program in Southern Belgium (Wallonia-Brussels Federation) where there is 59.000 newborns/year, among whom 6 are affected by spinal muscular atrophy.

ELIGIBILITY:
Inclusion Criteria:

* All newborns in southern Belgium

Exclusion Criteria:

* Newborns whose parents refuse screening

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns
Sampling Method: Non-Probability Sample
Enrollment: 136339 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Cases detected | march 2018-March 2021
  Number of cases detected, false negative and false positive cases

SECONDARY OUTCOMES:
Incidence of SMA | March 2018-March 2021
  to gather epidemiological data on SMA in Wallonia-Brussels Federation (carrier frequency, number of cases/year).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, PhD, Principal Investigator — CRMN
Locations (1):
- CRMN, Hôpital La Citadelle, Liège, Wallonia, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boemer F, Caberg JH, Dideberg V, Dardenne D, Bours V, Hiligsmann M, Dangouloff T, Servais L. Newborn screening for SMA in Southern Belgium. Neuromuscul Disord. 2019 May;29(5):343-349. doi: 10.1016/j.nmd.2019.02.003. Epub 2019 Feb 15. PMID 31030938